CLINICAL TRIAL: NCT06912165
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Study to Evaluate the Efficacy and Safety of WD-890 Tablets for the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: A Study of WD-890 in Participants With Moderate-to-Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Wenda Pharma Technology LTD. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WENDA890PSO-001
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Brief Description of Focus of Study

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: WD-890 Dose 1 QD and Placebo (Experimental)
  Interventions: Drug: WD-890 tablet
- Group 2: WD-890 Dose 2 QD and Placebo (Experimental)
  Interventions: Drug: WD-890 tablet
- Group 3: WD-890 Dose 3 QD and Placebo (Experimental)
  Interventions: Drug: WD-890 tablet
- Group 4: Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WD-890 tablet — Participants will receive WD-890 Dose 1 QD and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Arms: Group 1: WD-890 Dose 1 QD and Placebo
Drug: WD-890 tablet — Participants will receive WD-890 Dose 2 QD and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Arms: Group 2: WD-890 Dose 2 QD and Placebo
Drug: WD-890 tablet — Participants will receive WD-890 Dose 3 QD and placebo from Week 0 through Week 16. Participants will receive placebo to maintain the blinding of dose regimens.
  Arms: Group 3: WD-890 Dose 3 QD and Placebo
Drug: Placebo — Participants will receive placebo QD from Week 0 through Week 16.
  Arms: Group 4: Placebo

SUMMARY:
Th purpose of the study is to evaluate the dose response of WD-890 in efficacy at Week 16 in participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
The total duration of this study is up to 24 weeks which includes a screening period of less than or equal to (<=) 4 weeks, a 16-week treatment period, and a 4-week safety follow-up period. Aged 18 to 70 years (inclusive) were enrolled in this study. Participants were randomized to receive WD-890 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant aged 18 to 70 years(inclusive)at the time of informed consent.
* Diagnosis of plaque psoriasis for at least 6 months prior to the screening visit.

  ≥10% of BSA involvement at screening visit and randomization;
* Psoriasis Area and Severity Index (PASI) score ≥12 and static Physician's Global Assessment (sPGA) ≥3 at screening visit and randomization

Exclusion Criteria:

* Participant has a nonplaque form of psoriasis (for example, erythrodermic, guttate, inverse, pustular,or drug induced psoriasis.)
* Has uncontrolled arterial hypertension characterized by a systolic blood pressure (BP) ≥160 mm Hg or diastolic BP ≥100 mm Hg Note: Determined by 2 consecutive elevated readings. If an initial BP reading exceeds this limit, the BP may be repeated once after the subject has rested sitting for ≥10 minutes. If the repeat value is less than the criterion limits, the second value may be accepted
* Class III or IV congestive heart failure by New York Heart Association Criteria
* Participant with a history of chronic bacterial infections (e.g., chronic pyelonephritis, chronic bronchiectasis, or chronic osteomyelitis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 75 Score at Week 16 | Screening up to Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Skin Diseases, Institute of Dermatology, Chinese Academy of Medical Sciences, Peking Union Medical College, Nanjing, Jiangsu, China